CLINICAL TRIAL: NCT02875860
Title: TOTAL TRIAL: Randomized Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) Versus Expectant Management During Pregnancy in Fetuses With Left-Sided and Isolated Congenital Diaphragmatic Hernia and Moderate Pulmonary Hypoplasia
Brief Title: 'TOTAL' (Tracheal Occlusion To Accelerate Lung Growth) Trial
Acronym: TOTAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael A Belfort (Other)
Collaborators: Baylor College of Medicine (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor-Investigator, Michael A Belfort, Principal Investigator, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-39398
Record Dates: First submitted 2016-08-05; First posted 2016-08-23 (Estimated); Results first posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Hernia; Hernia, Diaphragmatic; Hernia, DIaphragmatic, Congenital; Pathological Conditions, Anatomical; Congenital Abnormalities; Congenital Diaphragmatic Hernia; Fetal Anomaly; Fetal Surgery; Pulmonary Hypoplasia
Keywords: CDH; Congenital Diaphragmatic Hernia; Fetal Tracheal Occlusion; FETO; plug-unplug; GoldBal2; Balloon; Goldvalve Balloon; TOTAL
MeSH Terms: conditions — Hernia; Hernia, Diaphragmatic; Pathological Conditions, Anatomical; Congenital Abnormalities; Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standardized postnatal care (Expectant) (Other): Mothers will be expectantly managed during pregnancies and babies receive standardized postnatal care at a tertiary center used to manage babies with CDH. The recommendation is that they adhere to consensus guidelines published on the study website.
  Interventions: Other: Standardized postnatal care
- Prenatal Intervention (FETO) (Experimental): Patients will undergo fetoscopic endoluminal tracheal occlusion and ideally prenatal reversal of the occlusion followed by standardized postnatal care as in the expectant . In this study FETO (where GoldBal2 detachable balloon and Baltaccidbpe100 Delivery Catheter are used) is to be done between 30 weeks plus 0 day and 31 weeks plus 6 days and removal of the balloon at 34 weeks plus 0 day to 34 weeks plus 6 days.
  Interventions: Device: GoldBal2 detachable balloon; Device: Baltaccidbpe100 Delivery Catheter; Other: Standardized postnatal care

INTERVENTIONS:
Device: GoldBal2 detachable balloon — Placement of the balloon using the plug/unplug method.
  Arms: Prenatal Intervention (FETO)
Device: Baltaccidbpe100 Delivery Catheter — The catheter assists with implanting the balloon in the plug/unplug method.
  Arms: Prenatal Intervention (FETO)
Other: Standardized postnatal care — After birth, the babies will receive standardized postnatal care at a tertiary center used to manage babies with CDH. The recommendation is that they adhere to consensus guidelines published on the study website. For detailed description on this please visit https://www.karger.com/Article/Abstract/320622

SUMMARY:
This trial will test whether temporary fetoscopic endoluminal tracheal occlusion (FETO) rather than expectant management during pregnancy, followed by standardized postnatal management, increases survival at discharge and decreases oxygen need at 6 months in case of survival till discharge.

DETAILED DESCRIPTION:
This is a multi-center, non-blinded randomized controlled trial in fetuses with isolated moderate CDH, i.e. moderate lung hypoplasia (as determined by prenatal assessment of lung development). It essentially compares fetal therapy added to conventional postnatal care, versus expectant prenatal management during pregnancy followed by conventional postnatal care.

Enrollment:

Following completion of an inclusion/exclusion criteria checklist and obtaining informed consent, the subject will be randomized into two groups ("FETO" and "expectant").

Procedures:

Group I: Standardized postnatal care (expectant group): mothers will be expectantly managed during pregnancies and babies receive standardized postnatal care at a tertiary center used to manage babies with CDH. The recommendation is that they adhere to consensus guidelines published on the study website.

Group II: Prenatal intervention (FETO group): patients will undergo fetoscopic tracheal occlusion and ideally prenatal reversal of the occlusion followed by standardized postnatal care as in I. In this study FETO is to be done between 30 weeks plus 0 day and 31 weeks plus 6 days and removal of the balloon at 34 weeks plus 0 day to 34 weeks plus 6 days.

This study trial is a pragmatical or efficacy trial: ideally mothers will deliver after removal of the balloon at those tertiary centers, typically offering postnatal care for the patient involved. In group II (FETO-group), mothers will, in between placement and removal of the balloon, thus carrying a fetus with obstructed airways, ideally remain under the care of our local fetal treatment center (further referred to as FETO center). As many as possible precautions are taken to avoid problems with balloon removal in case of earlier than expected delivery.

* Balloons are to be electively removed prior to 35 weeks. FETO centers will provide 24/24 hours and 7/7 days services for management of fetuses with obstructed airways, either in utero or during labor and delivery.
* Patients in the study and randomized to FETO, will be encouraged to stay near the FETO center. After reversal of the occlusion the patient will be referred to the tertiary care center where delivery and postnatal care will be undertaken. If the patient is not remaining at or close to the FETO center, the postnatal treatment center should organize likewise EXIT services.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or more, who are able to consent,
2. Singleton pregnancy,
3. Chromosomally normal fetus,
4. Gestation at randomization prior to 31 weeks plus 5 days or so that occlusion is done at the latest on 31 weeks plus 6 days,
5. Fetus is estimated to have moderate pulmonary hypoplasia, defined prenatally as:

   • O/E LHR 25-34.9% (included; irrespective of the position of the liver) • O/E LHR 35-44.9% (included) with intrathoracic liver herniation as determined by ultrasound or MRI.

   The O/E LHR will be determined by the FETO centers as follows:
   * Measurement of the contralateral lung area preferentially by the tracing method at the 4-chamber view of the heart; if by other method adjusted normative ranges must be used.
   * Measurement of the head circumference at the standard biparietal view of the head
   * The observed lung area: calculation of the LHR as the ratio of the measurements of the lung area to head circumference
   * The expected lung area is the lung area of a normal gestational age match, as determined by the head circumference of the index case in a normogram established for the same measurement method (tracing method in this case). A calculator for this will be available on the website of the study.
   * Calculation of the observed over expected lung area,
6. Acceptance of randomization and the consequences for the further management during pregnancy and thereafter, this includes the required observation following FETO surgery, which lasts up to 4 weeks after balloon is in place,
7. The patients must undertake the responsibility for either remaining close to, or at the FETO center, or being able to travel swiftly and within acceptable time interval to the FETO center until the balloon is removed. Intended postnatal treatment center must subscribe to suggested guidelines for "standardized postnatal treatment," and
8. Provide written consent to participate.
9. Fetus with no major anomalies that would impact the clinical course or outcomes.

Exclusion Criteria:

1. Maternal contraindication to fetoscopic surgery or severe medical condition in pregnancy that make fetal intervention risky,
2. Technical limitations precluding fetoscopic surgery, such as severe maternal obesity, uterine fibroids or potentially others, not anticipated at the time of writing this protocol,
3. Preterm labor, cervix shortened (<15 mm at randomization) or uterine anomaly strongly predisposing to preterm labor, placenta previa,
4. Patient age less than 18 years,
5. Psychosocial ineligibility, precluding consent,
6. Diaphragmatic hernia: right-sided or bilateral, major anomalies, isolated left-sided outside the O/E LHR limits for the inclusion criteria, and
7. Patient refusing randomization, to comply with required 4-week observation after balloon placement, or to comply with return to FETO center during the time period the airways are occluded or for elective removal of the balloon.
8. Patient allergic to latex.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Belfort, MD, PhD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Baylor College of Medicine/Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jani J, Nicolaides KH, Keller RL, Benachi A, Peralta CF, Favre R, Moreno O, Tibboel D, Lipitz S, Eggink A, Vaast P, Allegaert K, Harrison M, Deprest J; Antenatal-CDH-Registry Group. Observed to expected lung area to head circumference ratio in the prediction of survival in fetuses with isolated diaphragmatic hernia. Ultrasound Obstet Gynecol. 2007 Jul;30(1):67-71. doi: 10.1002/uog.4052. PMID 17587219
- [Background] Jani JC, Benachi A, Nicolaides KH, Allegaert K, Gratacos E, Mazkereth R, Matis J, Tibboel D, Van Heijst A, Storme L, Rousseau V, Greenough A, Deprest JA; Antenatal-CDH-Registry group. Prenatal prediction of neonatal morbidity in survivors with congenital diaphragmatic hernia: a multicenter study. Ultrasound Obstet Gynecol. 2009 Jan;33(1):64-9. doi: 10.1002/uog.6141. PMID 18844275
- [Background] Deprest J, Gratacos E, Nicolaides KH; FETO Task Group. Fetoscopic tracheal occlusion (FETO) for severe congenital diaphragmatic hernia: evolution of a technique and preliminary results. Ultrasound Obstet Gynecol. 2004 Aug;24(2):121-6. doi: 10.1002/uog.1711. PMID 15287047
- [Background] Jani J, Nicolaides K, Gratacos E, et al. 558: Short term neonatal morbidity in severe left-sided congenital diaphragmatic hernia treated by tracheal occlusion before 30 weeks. Am J Obstet Gynecol Dec;197(6),Supplement:S162.
- [Background] Jani JC, Nicolaides KH, Gratacos E, Vandecruys H, Deprest JA; FETO Task Group. Fetal lung-to-head ratio in the prediction of survival in severe left-sided diaphragmatic hernia treated by fetal endoscopic tracheal occlusion (FETO). Am J Obstet Gynecol. 2006 Dec;195(6):1646-50. doi: 10.1016/j.ajog.2006.04.004. Epub 2006 Jun 12. PMID 16769018
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Cannie MM, Jani JC, De Keyzer F, Allegaert K, Dymarkowski S, Deprest J. Evidence and patterns in lung response after fetal tracheal occlusion: clinical controlled study. Radiology. 2009 Aug;252(2):526-33. doi: 10.1148/radiol.2522081955. Epub 2009 Jun 9. PMID 19508989
- [Background] Reiss I, Schaible T, van den Hout L, Capolupo I, Allegaert K, van Heijst A, Gorett Silva M, Greenough A, Tibboel D; CDH EURO Consortium. Standardized postnatal management of infants with congenital diaphragmatic hernia in Europe: the CDH EURO Consortium consensus. Neonatology. 2010;98(4):354-64. doi: 10.1159/000320622. Epub 2010 Oct 27. PMID 20980772
- [Background] Snoek KG, Capolupo I, van Rosmalen J, Hout Lde J, Vijfhuize S, Greenough A, Wijnen RM, Tibboel D, Reiss IK; CDH EURO Consortium. Conventional Mechanical Ventilation Versus High-frequency Oscillatory Ventilation for Congenital Diaphragmatic Hernia: A Randomized Clinical Trial (The VICI-trial). Ann Surg. 2016 May;263(5):867-74. doi: 10.1097/SLA.0000000000001533. PMID 26692079
- [Background] Deprest JA, Flemmer AW, Gratacos E, Nicolaides K. Antenatal prediction of lung volume and in-utero treatment by fetal endoscopic tracheal occlusion in severe isolated congenital diaphragmatic hernia. Semin Fetal Neonatal Med. 2009 Feb;14(1):8-13. doi: 10.1016/j.siny.2008.08.010. Epub 2008 Oct 8. PMID 18845492
- [Background] Ruano R, Aubry MC, Barthe B, Mitanchez D, Dumez Y, Benachi A. Quantitative analysis of fetal pulmonary vasculature by 3-dimensional power Doppler ultrasonography in isolated congenital diaphragmatic hernia. Am J Obstet Gynecol. 2006 Dec;195(6):1720-8. doi: 10.1016/j.ajog.2006.05.010. Epub 2006 Jun 12. PMID 16769020
- [Background] Ostrea EM, Villanueva-Uy ET, Natarajan G, Uy HG. Persistent pulmonary hypertension of the newborn: pathogenesis, etiology, and management. Paediatr Drugs. 2006;8(3):179-88. doi: 10.2165/00148581-200608030-00004. PMID 16774297
- [Background] Congenital Diaphragmatic Hernia Study Group; Lally KP, Lally PA, Lasky RE, Tibboel D, Jaksic T, Wilson JM, Frenckner B, Van Meurs KP, Bohn DJ, Davis CF, Hirschl RB. Defect size determines survival in infants with congenital diaphragmatic hernia. Pediatrics. 2007 Sep;120(3):e651-7. doi: 10.1542/peds.2006-3040. PMID 17766505
- [Background] Gallot D, Boda C, Ughetto S, Perthus I, Robert-Gnansia E, Francannet C, Laurichesse-Delmas H, Jani J, Coste K, Deprest J, Labbe A, Sapin V, Lemery D. Prenatal detection and outcome of congenital diaphragmatic hernia: a French registry-based study. Ultrasound Obstet Gynecol. 2007 Mar;29(3):276-83. doi: 10.1002/uog.3863. PMID 17177265
- [Background] Deprest JA, Evrard VA, Verbeken EK, Perales AJ, Delaere PR, Lerut TE, Flageole H. Tracheal side effects of endoscopic balloon tracheal occlusion in the fetal lamb model. Eur J Obstet Gynecol Reprod Biol. 2000 Sep;92(1):119-26. doi: 10.1016/s0301-2115(00)00435-8. PMID 10986445
- [Background] Chiba T, Albanese CT, Farmer DL, Dowd CF, Filly RA, Machin GA, Harrison M. Balloon tracheal occlusion for congenital diaphragmatic hernia: experimental studies. J Pediatr Surg. 2000 Nov;35(11):1566-70. doi: 10.1053/jpsu.2000.18311. PMID 11083424
- See also: Information for the public and healthcare providers. — http://www.TOTALtrial.eu
- See also: Information for the public and healthcare providers. — http://www.euroCDH.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Started | 2 | 3
Completed | 2 | 2
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO) | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (2.1) | 32.3 (7.6) | 32.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 3 | 5
BMI [Mean (Standard Deviation); unit: kg/m²] | 21.5 (0.7) | 27.6 (1.8) | 25.2 (3.6)
Observed to Expected Lung to Head Ratio at Enrollment [Median (Full Range); unit: percentage] — The observed to expected lung to head ratio (O/E LHR) is calculated by taking the ratio of the lung area divided by the head circumference, compared to a reference value for the gestational age at the time of measurement.
  percentage | 35.5 [31 to 40] | 31 [29 to 35] | 31 [29 to 40]
Gestational Age at Delivery [Median (Full Range); unit: weeks] | 39.2 [39.0 to 39.4] | 39.0 [38.0 to 40.1] | 39.0 [38.0 to 40.1]
Liver Herniation present at Enrollment [Count of Participants; unit: Participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Neonate Survival at Discharge From Hospital
Description: The null hypothesis to be tested is that there is no difference in survival between fetuses managed expectantly during pregnancy versus those undergoing antenatal therapy (FETO).
Time Frame: At hospital discharge, an average of 1.5 months
Population: Intent to Treat Population (all participants assigned to Expectant management or FETO).
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 3
Participants | 1 | 3

2. Primary Outcome: Participants Requiring Supplemental Oxygen
Description: The number of survivors requiring supplemental oxygen at 6 months of age
Time Frame: At 6 months of age
Population: Intent to Treat Population (all participants assigned to Expectant management or FETO) of all subjects who survived to discharge from the hospital (primarly outcome #1).
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 1 | 3
Participants | 1 | 1

3. Secondary Outcome: Grade of Oxygen Dependency
Description: Measured as FiO2 (oxygen) amount required as a grade (0-III) with Grade 0 indicating the best outcome and Grade III indicating the worst outcome.
  Grade 0 = No Bronchopulmonary Dysplasia (BPD); Grade I = FiO2 21% or room air; Grade II = FiO2 22-29%; Grade III = FiO2 >29%, CPAP or mechanical ventilation.
Time Frame: at 6 months of age
Population: As-treated ('per protocol') analysis. 1 patient in the expectant management arm died and is excluded from this analysis. 1 patient from the FETO arm withdrew prior to receiving the FETO procedure and is excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 1 | 2
Participants
  0 = No Bronchopulmonary Dysplasia (BPD) | 0 | 1
  I = FiO2 21% or room air | 0 | 0
  II = FiO2 22-29% | 1 | 1
  III = FiO2 >29%, CPAP or mechanical ventilation | 0 | 0

4. Secondary Outcome: Occurrence of Severe Pulmonary Hypertension
Description: Occurrence of severe pulmonary hypertension in the neonatal period.
Time Frame: During the first 4 weeks of life (neonatal period).
Population: As-treated ('per protocol') analysis. 1 patient from the FETO arm withdrew prior to receiving the FETO procedure and is excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

5. Secondary Outcome: ECMO (Extracorporeal Membrane Oxygenation) Support
Description: Need for extracorporeal membrane oxygenation (ECMO) in the neonatal period
Time Frame: Neonatal period (during the first 4 weeks of life)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 2
Participants | 1 | 2

6. Secondary Outcome: CDH Defect Size
Description: Postnatal grade classification (A-D) using CDH study group standardized system with A being the smallest defects and D being the largest defects.
  A = Defect entirely surrounded by muscle; B = Small (<50%) portion of the chest wall devoid of diaphragm tissue; C = Large (>50%) portion of the chest wall devoid of diaphragm tissue; D = Complete or near complete absence of the diaphragm.
Time Frame: Measured in neonate at delivery by MRI and/or ultrasound
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 2
Participants
  A: Entirely surrounded by muscle | 0 | 0
  B: Small (<50%) portion of the chest wall devoid of diaphragm tissue | 0 | 1
  C: Large (>50%) portion of the chest wall devoid of diaphragm tissue | 2 | 1
  D: Complete or near complete absence of the diaphragm | 0 | 0

7. Secondary Outcome: Number of Days in the NICU
Description: Length of stay in the neonatal intensive care unit measured in days
Time Frame: At the time of discharge from the NICU, an average of 1.5 months
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 1 | 2
days | 39 | 53 [49 to 57]

8. Secondary Outcome: Ventilatory Support
Description: Length of time participants required ventilator support measured in days.
Time Frame: During the first 4 weeks of life (neonatal period)
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 1 | 2
days | 18 | 21 [15 to 27]

9. Secondary Outcome: Number of Subjects With Periventricular Leukomalacia (PVL)
Description: As measured by presence in medical record ≤ 2 months postnatally by ultrasound (yes/no)
Time Frame: During first 2 months of life
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

10. Secondary Outcome: Neonatal Sepsis
Description: As measured by presence in medical record
Time Frame: During the first 4 weeks of life (neonatal period)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

11. Secondary Outcome: Intraventricular Hemorrhage
Description: Measured as presence in neonate during first month by MRI and/or ultrasound.
Time Frame: During first month of life
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

12. Secondary Outcome: Retinopathy of Prematurity
Description: Postnatal grade classification presence of grade III or higher using standardized system (yes/no)
Time Frame: At the time of discharge from the NICU, an average of 1.5 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

13. Secondary Outcome: Days to Full Enteral Feeding
Description: The number of days until full enteral feeding
Time Frame: At hospital discharge, an average of 1.5 months
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 1 | 2
days | 27 | 29.5 [23 to 36]

14. Secondary Outcome: Gastroesophageal Reflux
Description: Presence of reflux above 1/3 of esophagus on clinically indicated radiologic exam
Time Frame: At the time of discharge from the NICU, an average of 1.5 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 1 | 2
Participants | 1 | 0

15. Secondary Outcome: CDH (Congenital Diaphragmatic Hernia) Surgery Repair
Description: How many days from birth until the surgery is performed to repair the defect.
Time Frame: From the time of birth until discharge from the NICU
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 2
days | 1 [1 to 1] | 2.5 [2 to 3]

16. Secondary Outcome: Use of Patch in CDH Repair
Description: The number of participants who had a patch used in the repair of the CDH defect.
Time Frame: At the time of the surgical repair postnatally, up to 3 days postnatal
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

17. Secondary Outcome: Survival
Description: The number of participants that survived to 24 months of age
Time Frame: At 24 months of age
Population: Intent to Treat Population (all participants assigned to Expectant management or FETO).
Measure: Count of Participants; unit: Participants
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
Number analyzed (Participants) | 2 | 3
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the time period starting with enrollment of the first participant through 2 years post delivery of the baby.
Description: The deaths reported in All-Cause Mortality reflect neonates who died during the study.
Arm/Group | Standardized Postnatal Care (Expectant) | Prenatal Intervention (FETO)
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT02875860/Prot_SAP_000.pdf